CLINICAL TRIAL: NCT02486289
Title: A Randomized, Placebo-controlled Study to Explore Safety, Dose and Efficacy of NBMI in a Mercury Intoxicated Population
Brief Title: Pilot Proof of Concept Study of NBMI Treatment of Mercury Intoxication
Acronym: NBMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EmeraMed (Industry)
Collaborators: NBMI Science AB (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTI002
Record Dates: First submitted 2015-06-24; First posted 2015-07-01 (Estimated); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Mercury Poisoning
Keywords: Mercury toxicity poisoning
MeSH Terms: conditions — Mercury Poisoning | interventions — N,N'-Bis(2-mercaptoethyl)isophthalamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- NBMI (Emeramide) 100mg (Experimental): NBMI oral capsules 100mg administered once daily. Double dummy used for blinding i.e. 2 x 50mg NBMI + 1 x 200mg placebo capsule equals in total 3 capsules administered daily.
  Interventions: Drug: Emeramide
- NBMI (Emeramide) 300mg (Experimental): NBMI oral capsules 300mg administered once daily. Double dummy used for blinding i.e. 2 x 50mg NBMI + 1 x 200mg NBMI capsule equals in total 3 capsules administered daily.
  Interventions: Drug: Emeramide
- Placebo (Placebo Comparator): Placebo oral capsules administered once daily. Double dummy used for blinding i.e. 2 x 50mg size + 1 x 200mg size placebo capsules equal in total 3 capsules administered daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Emeramide — Mercury chelator NBMI ((N1,N3-bis(2-mercaptoethyl) isophthalamide)
  Other Names: NBMI; Irminix
  Arms: NBMI (Emeramide) 100mg; NBMI (Emeramide) 300mg
Drug: Placebo — NBMI Placebo
  Arms: Placebo

SUMMARY:
A randomized, placebo controlled, double blind proof of concept study of NBMI in treatment of mercury intoxication.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate the efficacy and safety of two doses of NBMI compared to placebo in mercury intoxicated patients.

ELIGIBILITY:
Inclusion criteria

1. Male or female subjects, age between 18 and 65 years, inclusive.
2. Urine-Hg ≥ 15 μg/L.
3. Mercury intoxication medical score sum (Doering et al. 2014) ≥ 5 or medical score sum ≥ 3 in combination with at least two of the following symptoms; social nervousness/withdrawal, irritability, memory loss, metallic taste, mental- and physical fatigue.
4. Has signed informed consent for participation.
5. Willingness and ability to comply with study procedures, visit schedules, and other instructions regarding the study.

Exclusion criteria

1. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subjects at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. Known or a medical history of renal disorder, significant renal failure, or high risk of renal failure.
3. Any clinically significant abnormalities in clinical chemistry or haematology results at the time of screening as judged by the investigator.
4. Known or suspected neurodegenerative disorder including but not limited to stroke, polio, Parkinson's and Alzheimer's disease.
5. Known or suspected drug or alcohol abuse.
6. Positive pregnancy test in women.
7. Serious bacterial and chronic viral infection such as human immunodeficiency virus (HIV) or hepatitis virus.
8. History of severe allergy/hypersensitivity or on-going allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to NBMI.
9. History of allergy/hypersensitivity to bisulphites (e.g. red/white wine).
10. Participation in any other clinical study that included drug treatment within three months of the first administration of investigational product.
11. Use of other therapies for mercury intoxication including metal chelators within three months.
12. Investigator considers subject unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Mercury Intoxication Medical Score Sum | 45 days
  Changes from baseline in mercury intoxication medical score sum compared between treatment arms.

SECONDARY OUTCOMES:
Individual components of Mercury Intoxication Medical Score Sum | 45 days
  Changes from baseline in individual components of the mercury intoxication medical score sum compared between treatment arms.
Fatigue score | 15 days
  Changes from baseline in fatigues score sum compared between treatment arms.
Neuromotoric functions | 45 days
  Changes from baseline in neuromotoric functions objectively assessed and quantified using computerized systems such as CATSYS compared between treatment arms.
Blood mercury levels | 45 days
  Changes from baseline in blood mercury level compared between treatment arms.
Urine mercury levels | 45 days
  Changes from baseline in urine mercury level compared between treatment arms.
NBMI blood levels | 14 days
  NBMI blood levels 0-24 hours after the first and last dose (day 14 dose)
NBMI urine levels | 14 days
  NBMI urine levels 0-24 hours after the first and last dose (day 14 dose)
Adverse events | 45 days
  Adverse event frequency, type and severity compared between treatment arms.
Safety laboratory assessments | 45 days
  Changes from baseline in clinical chemistry and haematology tests compared between treatment arms.
Vital signs | 45 days
  Changes from baseline in vital signs compared between treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Augusto Focil Baquerizo, MD, Principal Investigator — FOMAT Medical Research
Locations (1):
- Hospital Doctor Humberto Molina, Zaruma, Ecuador

REFERENCES:
- [Derived] Schutzmeier P, Focil Baquerizo A, Castillo-Tandazo W, Focil N, Bose-O'Reilly S. Efficacy of N,N'bis-(2-mercaptoethyl) isophthalamide on mercury intoxication: a randomized controlled trial. Environ Health. 2018 Feb 14;17(1):15. doi: 10.1186/s12940-018-0358-1. PMID 29444690